CLINICAL TRIAL: NCT05514899
Title: Effects of Cannabidiol and Tetrahydrocannabinol on the Microbiome, Endocannabinoids, and Neuroinflammation in HIV
Brief Title: Effects of Cannabidiol and Tetrahydrocannabinol on Microbiome and Neuroinflammation in HIV
Acronym: CAMI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Ronald Ellis, Principal Investigator, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 802514
Record Dates: First submitted 2022-08-22; First posted 2022-08-25 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: HIV; Cannabis; THC; Neuroinflammatory Disease; Neuroinflammatory Response; Microbiome
MeSH Terms: conditions — Marijuana Abuse; Neuroinflammatory Diseases | interventions — Dronabinol; Cannabidiol

STUDY DESIGN:
Intervention Model Description: This will be a double-blind, randomized, 2-sequence crossover trial of CBD versus THC to reduce systemic and neuro-inflammation. This design was chosen to balance consideration of addressing the key scientific questions (effects of CBD versus THC on the microbiome, ECS and inflammation and their interaction with HIV infection), scientific rigor, power and feasibility.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- THC first, then CBD (Experimental): THC 10mg daily for 2 weeks, followed by washout for 2 weeks, followed by CBD 600mg daily for 2 weeks
  Interventions: Drug: THC; Drug: CBD
- CBD first, then THC (Active Comparator): CBD 600mg daily for 2 weeks, followed by washout for 2 weeks, followed by THC 10mg daily for 2 weeks
  Interventions: Drug: THC; Drug: CBD

INTERVENTIONS:
Drug: THC — THC capsule
  Other Names: Delta-9 tetrahydrocannabinol; Tetrahydrocannabinol; Delta9-THC
Drug: CBD — oral solution
  Other Names: Cannabidiol

SUMMARY:
This study has the potential to contribute to a more complete understanding of the independent and combined effects of cannabis use and HIV on the brain and on inflammation. Such knowledge may inform future strategies for treating brain disease and inflammation. Participants will be randomly assigned to one of two groups, both of which will receive the same treatment in a different order over a period of about 6 weeks. The visits include physical examinations, blood tests, and other procedures designed to monitor subject safety and measure the effects of the study drug.

DETAILED DESCRIPTION:
This project will characterize the microbiome and endocannabinoid system (ECS) in people with HIV (PWH) and how they relate to neuroinflammation and blood-brain barrier (BBB) function. The study hypothesizes that pathogenic alterations in the gut microbiota (dysbiosis) and impaired gut barrier integrity (leaky gut) are mediators between the ECS, neuroinflammation and BBB dysfunction in HIV. The major goals are to (1) characterize the gut microbiota and ECS in response to exogenous cannabinoid exposure in both PWH and people without HIV (PWoH); (2) characterize patterns of HIV-associated inflammation (innate, adaptive, T-cell, B-cell) in blood and cerebrospinal fluid (CSF) in response to controlled cannabis exposure; (3) assess effects of cannabinoid exposure on these patterns and how they are mediated through changes in the ECS, gut microbiota and gut barrier function. The investigators will perform a clinical trial of 50 PWH and 50 PWoH exposed in a randomized, cross-over fashion to 14 days each of oral THC and CBD to determine if treatment with either phytocannabinoid reduces inflammation and improves gut function. The experimental approach will use fecal shotgun metagenomic sequencing to characterize the gut microbiome, with particular attention to aerotolerant bacteria, pro-inflammatory species, Prevotella spp., Bifidobacterium and Bacteroides spp. and butyrate-producing bacteria. We will evaluate how the microbiota and leaky gut relate to neuroinflammation and impaired BBB function, the latter potentially leading to increased central nervous system (CNS) exposure to microbially-produced pro-inflammatory ligands. The rationale for the study is that virologic suppression on antiretroviral therapy (ART) does not normalize gut lymphoid tissue cluster of differentiation 4 (CD4)+ T cell depletion, leaky gut, dysbiosis, chronic gut inflammation, and microbial antigen translocation (MAT). These alterations ultimately drive systemic and CNS inflammation. Compromised gut barrier function due to altered tight junctions, apoptosis and reduced epithelial cell proliferation and repair render PWH susceptible to increased tissue exposure to pro-inflammatory ligands produced by gut microbiota and are important in HIV neuropathogenesis. Of particular relevance here are recent findings that the ECS in the large intestine interacts with the gut microbiota to regulate epithelial barrier permeability. Thus, constituents of cannabis, acting through the EC systems in the gut, brain and immune system, may be therapeutic. The existing literature suggests that the two principal constituents of cannabis, Δ9-tetrahydrocannabinol (THC) and cannabidiol (CBD), have differential effects on the ECS.

ELIGIBILITY:
1. Aged 21 to 70 years old
2. Possess the capacity to provide informed consent to a set of neuromedical assessment procedures.
3. Experience with cannabis use at least once in the past 5 years without major adverse effects (e.g., psychosis, syncope)
4. No or low cannabis use in the past 2 weeks, defined as no cannabis exposure or use or use limited to only once in the past 2 weeks.
5. Willing to abstain from use of cannabis, CBD, THC, or synthetic cannabinoids outside the study during the 6-week intervention
6. Individuals with HIV must meet the following criteria

   1. Virally suppressed on stable ART for at least 6 months and have no more than 1 prior event of virologic failure (i.e., required change in ARTs due to virologic failure)
   2. Stage 1 or 2 infection
   3. Have a "normal" CD4 count defined as ≥350 cells/microliter
   4. No significant history of ART regimen adherence challenges
7. Ability to adhere to the study visit schedule.

Exclusion Criteria:

1. Exclusion criteria will be: any substance use disorder (abuse or dependence) other than cannabis in the last 30 days;
2. Significant cognitive impairment such as Dementia, including Alzheimer's disease
3. Pregnancy or lactation, or unwillingness to prevent pregnancy during the trial; refusal to maintain highly effective contraceptive methods (e.g., implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), sexual abstinence or vasectomized partner) during the study for persons of child-bearing potential or those with partners of child-bearing potential
4. Evidence of moderately or worse compromised liver or kidney function, including moderate (Child-Hugh B) or severe (Child-Hugh C) hepatic impairment and AST and ALT above ULN and total bilirubin above ULN;
5. Evidence of significant cardiovascular risk, resting heart rate <50 or >110 beats per minute, uncontrolled hypertension (systolic blood pressure <80 or >140 mmHg; diastolic blood pressure <50 or >90 mmHg), history of myocardial infarction, congestive heart failure, or arrhythmia);
6. Evidence of chronic pulmonary disease requiring supplemental oxygen;
7. Active, recent, or remote medical history of hepatobiliary-related illness, including elevated transaminase levels above 3 times the upper limit of normal accompanied by elevations in total bilirubin above 2 times the upper limit of normal at screening;
8. Insulin dependent diabetics
9. Allergy to the study drugs or any of their constituents including sesame
10. Use of medications with absolute contraindicated or potential significant interactions
11. Use of sedating medications
12. Weighing less than 60 kg at screening to minimize the risk of elevated transaminases as a result of exposure to cannabidiol;
13. Active, uncontrolled psychiatric disorder with psychotic features, severe depression, or suicidality; Participants will be excluded if they have had a history of suicide attempt, recent suicidal ideation or behavior as indexed by their Beck Depression Inventory-II (BDI-II) score is greater than or equal to 29 (severe depression).
14. Neurologic disorder that could compromise interpretation of study findings, including uncontrolled seizure disorder (active seizures within the past 3 months), multiple sclerosis, Parkinson's disease, Alzheimer's disease, and recent (past 3 months) cerebral infarction or hemorrhage with neurological sequelae.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
PC1 | Change from baseline to Week 2
  A composite marker of inflammation, comprising the first component (PC1, a unitless measure) of the principal component analysis (PCA) of 7 soluble biomarkers in blood (soluble CD163 [sCD163], interferon gamma [IFN-gamma], interleukin 6 [IL-6], C-reactive protein [CRP], CC motif chemokine ligand 2 [CCL2], neopterin and soluble tumor necrosis factor - type II [sTNFRII]), all measured in picograms/milliliter
PC1 | Change from Week 4 to Week 6
  A composite marker of inflammation, comprising the first component (PC1, a unitless measure) of the principal component analysis (PCA) of 7 soluble biomarkers in blood (soluble CD163 [sCD163], interferon gamma [IFN-gamma], interleukin 6 [IL-6], C-reactive protein [CRP], CC motif chemokine ligand 2 [CCL2], neopterin and soluble tumor necrosis factor - type II [sTNFRII]), measured in picograms/milliliter

SECONDARY OUTCOMES:
blood-brain barrier (BBB) | Change from baseline to Week 2
  BBB markers: claudin, suPAR, CSF/serum albumin ratio, MMP-2, occludin, all measured in picograms/milliliter
blood-brain barrier (BBB) | Change from Week 4 to Week 6
  BBB markers: claudin, suPAR, CSF/serum albumin ratio, MMP-2, occludin, measured in picograms/milliliter

CONTACTS AND LOCATIONS:
Overall Officials: Ronald J Ellis, MD, PhD, Principal Investigator — UC San Diego
Locations (1):
- HIV Neurobehavioral Research Program (HNRP), San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
Data sharing will be considered upon request